CLINICAL TRIAL: NCT03393845
Title: A Phase II Study of Pembrolizumab Plus Fulvestrant in Hormone Receptor Positive, HER-2 Negative Advanced/Metastatic Breast Cancer Patients: Big Ten Cancer Research Consortium BTCRC-BRE16-042
Brief Title: Study of Pembrolizumab Plus Fulvestrant in Hormone Receptor Positive, HER-2 Negative Advanced/Metastatic Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Chan, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Nancy Chan, MD, Sponsor Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-BRE16-042
Record Dates: First submitted 2018-01-02; First posted 2018-01-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Fulvestrant (Experimental): Pembrolizumab 200m IV q3W + Fulvestrant. Loading dose 500mg IV IM q2W x3 followed by 500mg IM q4W
  Interventions: Drug: Pembrolizumab; Drug: Fulvestrant

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg IV, 21 day cycles
  Other Names: Keytruda
Drug: Fulvestrant — Fulvestrant, 500mg IM, Loading dose: C1 D1 & 15. Thereafter, Q4 wks
  Other Names: Faslodex

SUMMARY:
Pembrolizumab Plus Fulvestrant in Hormone Receptor Positive, HER-2 Negative Advanced/Metastatic Breast Cancer Patients

DETAILED DESCRIPTION:
This is a non-randomized, multi-site, open-label Phase II trial for subjects with metastatic, hormone receptor positive, HER2 negative breast cancer. The study will enroll 47 patients to evaluate the anti-tumor activity of pembrolizumab with fulvestrant as measured by RECIST 1.1 tumor response and by progression free survival. We expect that if the immune response is augmented by the addition of pembrolizumab, significant change in durability of response will be noted.

Patients will be treated with pembrolizumab dosed at 200 mg intravenous infusion in combination with standard fulvestrant 500mg intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Men [29] and women ≥ 18 years of age at the time of informed consent. NOTE: Both pre- and post-menopausal women are eligible. Patients who are premenopausal should either undergo bilateral oophorectomy or receive ovarian suppression according to institutional standards. Male patients will be treated as premenopausal females and receive a GnRH agonist.
* ECOG Performance Status of 0 or 1 within 28 days prior to registration.
* Histologic or cytologic diagnosis of metastatic breast cancer.
* Has received no more than two lines of prior therapy for advanced non-resectable/metastatic disease. Prior lines can can be either chemotherapy or hormonal therapy. Prior or current fulvestrant is allowed. Combination therapy is considered as one regimen.
* Tumor is estrogen receptor positive (ER+) and/or (PR+), HER-2 negative (HER2-). ER and PR positivity is defined as >1%. HER-2 negative is defined as by IHC (0, 1+) or FISH. HER2 positive test result includes: Single-probe average HER2 copy number ≥6.0 signals/cell; Dual-probe HER2/CEP17 ratio ≥2.0 with an average HER2; copy number ≥4.0 signals/cell; Dual-probe HER2/CEP17 ratio ≥2.0 with an average HER2copy number <4.0 signals/cell; or Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number ≥6.0 signals/cell. Equivocal findings for IHC as 2+ should be reflexed to FISH. Equivocal results by FISH may be considered with approval from the Sponsor-Investigator.
* Measurable disease based on RECIST 1.1 within 28 days prior to registration. Except in patients with bone-only disease, in the absence of measurable disease, evaluable bone lesion is allowed. NOTE: Bone-only disease is the sole non-measurable disease site allowed and biopsy is required. Measurable disease is required in all other cases.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. NOTE: Subjects for whom newly-obtained fresh tissue samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor-Investigator.
* Normal cardiac function as determined by treating physician per institutional standards via echocardiogram (ECHO) performed within 28 days prior to registration.
* Prior chemotherapy must be completed at least 28 days prior to registration or at least 14 days prior to registration for targeted therapy.
* Prior hormonal therapy or radiation therapy must be completed at least 14 days prior to registration. If subject is currently receiving fulvestrant, it may continue without interruption as per standard of care.
* The subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or baseline. NOTE: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. NOTE: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to study registration, as determined by the enrolling physician.
* Demonstrate adequate organ function as defined in the table below; all screening labs will be performed within 28 days of study registration.

  * Hematological

    * Absolute Neutrophil Count (ANC): ≥ 1500/mm3
    * Platelets: ≥100,000 / mcL
    * Hemoglobin (Hgb): ≥ 9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Renal

    ---Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤1.5 × upper limit of normal (ULN) OR ≥30 mL/min for subjects with creatinine levels > 1.5 × institutional ULN
  * Hepatic

    * Serum total bilirubin: ≤ 1.5 X ULN OR
    * Direct bilirubin ≤ ULN for subjects with total bilirubin levels: > 1.5 ULN
    * AST (SGOT) and ALT (SGPT): ≤ 2.5 × ULN
    * Albumin: >2.5 mg/dL
  * Coagulation ---International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT): ≤1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance will be calculated per institutional standard.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to study registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: Females are considered of childbearing potential unless: they are postmenopausal; are surgically sterile; or they have a congenital or acquired condition that prevents childbearing. See the protocol for definitions. NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Females and males of reproductive potential must be willing to abstain from heterosexual activity which could result in pregnancy or agree to use an adequate method of contraception as outlined in the protocol. Hormonal contraceptives are contraindicated in this population and are not allowed. Contraception will begin from the time of informed consent through 120 days after the last dose of study drug(s).

Exclusion Criteria:

* Is currently receiving an investigational agent or has received an investigational agent or used an investigational device within 28 days of study registration.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.

NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Has a known history of active TB (Bacillus Tuberculosis). NOTE: TB testing is not required.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). NOTE: HIV testing is not required.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

NOTE: Hepatitis B and Hepatitis C testing is not required.

* Hypersensitivity to pembrolizumab or any of its excipients.
* Has received prior chemotherapy within 28 days prior to study registration or has received prior hormonal/targeted therapy within 14 days prior to study registration
* More than two lines of chemotherapy or more than two lines of hormonal therapy excludes participation.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has known history of non-infectious pneumonitis/interstitial lung disease that required steroids or has any evidence of active pneumonitis/interstitial lung disease.
* Has known history of, or any evidence of active interstitial lung disease, Class II-IV congestive heart failure, or myocardial infarction within 6 months from randomization.
* Active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Breastfeeding during the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has received a live vaccine or live-attenuated vaccine within 30 days of study registration. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Ratio (CBR) | 36 months
  Clinical benefit ratio (CBR) is defined as the percentage of patients that achieve CR, PR, or stable disease for a minimum of four months. Patients will be evaluated for response by RECIST 1.1 and irRECIST.

SECONDARY OUTCOMES:
Safety profile of pembrolizumab plus fulvestrant | 36 months
  To describe the toxicity profile of pembrolizumab plus fulvestrant in patients with hormone receptor positive, HER2 negative advanced/metastatic breast cancer. The toxicity profile will report all grade 3 and 4 toxicities as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4
Progression free survival (PFS) | 36 months
  Progression free survival is defined as the time from date of treatment start until the criteria for disease progression is met or death from any cause. PFS will be assessed by RECIST 1.1 and irRECIST
Durable response rate (DRR) | 36 months
  Durable response rate is defined as the number of months that a stable disease, partial or complete response is observed.
Overall Survival | 36 months
  Overall survival is defined as defined as the time from date of treatment start until death

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chan, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Michigan State University, Breslin Cancer Center, Lansing, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Clinical Cancer Center, New York, New York
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided